CLINICAL TRIAL: NCT03624244
Title: Randomized Comparative Prospective Multicentre Phase II Trial Evaluating Clinical Impact of Interruption VS Maintenance of AI in Patients with Locally Advanced/ Metastatic LGESS
Brief Title: Evaluation of Clinical Impact of Interruption VS Maintenance of AI in Patients with Locally Advanced/ Metastatic Low Grade Endometrial Stromal Sarcoma (LGESS)
Acronym: BFR-ESS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET17-200 BRF-ESS
Record Dates: First submitted 2018-07-18; First posted 2018-08-10 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Low Grade Endometrial Stromal Sarcoma
Keywords: Low Grade Endometrial Stromal Sarcoma; Aromatase inhibitors
MeSH Terms: conditions — Endometrial Stromal Tumors | interventions — Aromatase Inhibitors; Anastrozole; exemestane; Letrozole

STUDY DESIGN:
Intervention Model Description: Phase II comparative multicentre prospective randomised (1:1 ratio) open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interruption of aromatase inhibitors (Experimental): Interruption of aromatase inhibitors until progression disease. At disease progression, AI can be reintroduced.
  Interventions: Drug: Aromatase Inhibitors
- Maintenance of aromatase inhibitors (Other): Maintenance of aromatase inhibitors
  Interventions: Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Aromatase Inhibitors — Maintenance of AI versus interruption of AI
  Other Names: ANASTRAZOLE, ARIMIDEX, AROMASINE, EXEMESTANE, FEMARA, LETROZOLE

SUMMARY:
The primary objective is to compare the progression-free survival (PFS) between aromatase inhibitors interruption and aromatase inhibitors maintenance strategies in patients with a locally advanced or metastatic Low Grade Endometrial Stromal Sarcoma (LGESS).

DETAILED DESCRIPTION:
Uterine sarcomas are rare tumors with an incidence of 1.7/100 000 women per year, including 20% of endometrial stromal sarcomas (ESS). Patients with low grade ESS (LGESS) have a good prognosis with a 5-year overall survival rates ranging from 66 to 98%, depending on the stage of the disease.

Majority of LGESS report estrogen receptor (ER) and/or progesterone receptor positive and a chromosomal translocation with JAZF1-SUZ12.

Based on the current European Society of Medical Oncology (ESMO)guidelines, the standard treatment for patients with early/non metastatic ESS is total hysterectomy plus or less bilateral salpingo-oophorectomy. The use of hormonal therapy (HT) for advanced or metastatic disease is recommended based on retrospective data from small series providing evidence that HT have an anti-tumor activity on LGESS. HT includes aromatase inhibitors (AI), progestins and gonadotrophin-releasing hormone.

Very few data are available in this rare disease, but retrospective analyses show that AI may provide response rates of 46 to 67% in metastatic LGESS patients (7% complete response, 60% partial response), with a mean duration of response of 24 months.

Even if AI are effective and well tolerated, chronical mild to moderate (grade 1-2) side-effects (arthritis, hot-flashes, osteoporosis, hypercholesterolemia, cardiac events) have a negative impact on patient's well-being because of the treatment long term duration and need to be balanced in such long term survival.

To date, the question of the optimal duration of HT in LGESS is still pending. The investigator propose an open-label, randomized, multicenter phase II study aiming at determining the feasibility of interruption of AI in patients with locally advanced or metastatic LGESS after long term stabilization or response to AI. The study will use a sequential bayesian design allowing for continuous monitoring of the main efficacy outcome, thus leading to a smaller more informative trial, and specifically tied to decision making. This design is particularly suited to characterize efficacy signals in the context of a very rare pathology. Moreover JAZF1-JJAZ1 fusion gene is not identified in all LGESS.

Ancillary studies will provide precious data aiming at:

* Identifying predictive factors of prolonged response to HT or late resistance (Next Generation Sequencing and Comparative Genome Hybridization).
* Evaluating sociobehavioral (only for French sites) of patients by following questionnaire: Zimbardo Time Perspective Inventory (ZTPI) , Functional, Communicative and Critical Health Literacy/ 14-item Health Literacy Scale (FCCHL/HLS14), VICAN, Fear of Cancer Recurrence (FCR) and Patient-Generated Index (PGI).

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years;
* Histological confirmation of low grade ESS;
* Locally advanced or metastatic disease at diagnosis or patient experiencing a tumor effraction during hysterectomy;
* Treatment with aromatase inhibitors (Anastrozole or Exemestane or Letrozole ) initiated either: for at least 24 months (in patients with no residual disease or non-measurable disease at the last AI initiation) OR for at least 36 months (in patients with measurable disease at the last AI initiation);
* Disease must be controlled at the time of the randomisation (objective response or stable disease) by the aromatase inhibitor initiated either for at least 24 or 36 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
* Covered by a medical insurance;
* Signed informed consent prior to any study-specific procedure.

Exclusion Criteria:

* Pregnant or breastfeeding woman;
* Patient concurrently using other approved or investigational antineoplastic agents;
* Major concurrent disease affecting cardiovascular system, liver, kidneys, hematopoietic system or else considered as clinically important by the investigator and that could be incompatible with patient's participation in this trial or would likely interfere with study procedures or results;
* Prior history of malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 3 years;
* Patients using prohibited concomitant and/or concurrent medications
* Contra-indication according to SmPCs.
* Patient requiring tutorship or curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression free survival

SECONDARY OUTCOMES:
Overall survival | From date of randomization to death due to any cause, assessed up to 60 months
  Overall survival
Time to first subsequent chemotherapy/treatment or death | From date of randomization to the earliest date of chemotherapy/treatment start date following study treatment discontinuation, or death due to any cause, whichever came first, assessed up to 60 months
  Time to first subsequent chemotherapy/treatment or death
Objective response rate after reintroduction of AI in the experimental arm | From the date of AI reintroduction in the experimental arm to the date of subsequent progression or date of death due to any cause, whichever came first, assessed up to 60 months
  Proportion of patients with a best overall response of Partial Response (PR) or Complete Response (CR) after AI reintroduction in the experimental arm
Progression free survival after reintroduction of AI in the experimental arm | From the date of AI reintroduction in the experimental arm to the date of subsequent progression or date of death due to any cause, whichever came first, assessed up to 60 months
  Progression free survival after reintroduction of AI in the experimental arm
Duration of response to AI after reintroduction | From the date of first objective response following the reintroduction of AI to the date of the first subsequent documented radiological progression or death due to any cause, whichever came first, assessed up to 60 months
  Duration of response to AI after reintroduction
Incidence of Treatment-Emergent Adverse Events | From date of randomization to follow-up visit Month 36 or death due to any cause, whichever came first, assessed up to 60 months
  Safety and Tolerability assessed according to the NCI-CTC AE version 5
Quality of Life using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) | Every 6 months until the 36th month for each patient
  Quality of Life using EORTC QLQ-C30 questionnaire. 64 questions related to cancer impact on health and daily activities composed this questionnaire. Each item has to be graded from 1 to 4 ( 1 = not at all; 4 = very much). More the score is high, worst the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAY-COQUARD, MD PhD, Principal Investigator — Centre Leon Berard
Locations (21):
- France (21):
  - CHU Besançon, Besançon
  - Insitut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Hopital La Timone, Marseille
  - Institut Paoli Calmette, Marseille
  - Institut de Cancérologie de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Pitié Salpétrière, Paris
  - AP-HP Hopîtal Cochin, Paris
  - Insitut Curie, Paris
  - Institut Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Hopital Privé de la Loire, Saint-Etienne
  - ICO Centre René Gauducheau, Saint-Herblain
  - CHUSE, Saint-Priest-en-Jarez
  - CHU Tours, Tours
  - Institut Gustave Roussy, Villejuif